CLINICAL TRIAL: NCT01471392
Title: Identigene STD Test Collection Kit Validation Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Identigene (Industry)
Collaborators: CRI Lifetree Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IDTG-100
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Infection
Keywords: Identigene; STD Test; Chlamydia; Gonorrhoeae; APTIMA; Sexually Transmitted Disease
MeSH Terms: conditions — Infections; Chlamydia Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Identigene STD Test Kit Arm (Experimental): Single-Arm trial where the group will complete the Identigene STD Test Kit at home and these results will be compared with the results from testing in the clinic with the Gen-Probe APTIMA kit. The subject will only be informed of the results from the approved test (Gen-Probe APTIMA) that is done in the clinic.
  Interventions: Device: STD Diagnostic Kit (Identigene)

INTERVENTIONS:
Device: STD Diagnostic Kit (Identigene) — The Identigene STD Test Collection Kit is an at-home kit that allows individuals to utilize the Gen-Probe technology to test for CT and NG in privacy and in a more convenient manner. The primary technology is the approved Gen-Probe APTIMA Combo 2 assay, which is repackaged into the Identigene kit for use by consumers. As such, the laboratory technology and testing method is identical to that of the Gen-Probe APTIMA Combo 2 assay, which has been cleared for in vitro diagnostic use.
  Other Names: Identigene STD Test Collection Kit

SUMMARY:
The overall goal of the present study is to provide evidence of concordant test results using the Identigene STD Test Collection Kit for self-collection and transport of specimens to a qualified testing laboratory. It is expected that this method will aid in detection of CT and NG and that offering a method of self-collection of a male urine or female vaginal swab specimen will encourage testing for CT and NG and improve the overall detection of reporting of these STDs by allowing persons who suspect they have the infection to be tested in a discrete and confidential manner. The reporting of CT and NG are underestimated and many subjects will not visit a clinic or obtain treatment if gone undetected. Thus, allowing a self-collection kit that is more convenient may result in improved reporting, identification of CT and NG positive individuals, and subsequent treatment to help prevent the spread of these diseases.

The purpose of this study is to demonstrate that the Identigene STD Test Collection Kit and labeled instructions for use instructions provide test results that are concordant (at least 95% or better) with test results obtained using the Gen-Probe APTIMA Combo 2 specimen collection and transport methods performed under the supervision of a healthcare provider. The laboratory technology and test method used for the IDTG-100.

DETAILED DESCRIPTION:
This is a multicenter study involving asymptomatic and symptomatic subjects who are at risk or suspect possible exposure to CT and/or NG. Approximately five (5) clinics will participate in the study. The clinics selected will be located in diverse geographical regions in order to represent populations with both high and low incidences of CT and NG and to represent different extremes in climate. The initial phase of the study enrolled approximately 500 qualifying subjects. An interim analysis was performed to determine whether changes in the study protocol were necessary. Changes to the protocol were identified and are incorporated in this amendment (amendment 4) of the study protocol. Specifically, males in the study will still collect urine specimens whereas women will now self-collect a vaginal swab specimen. Study subjects will only undergo one clinic visit rather than two as indicated in prior versions of the study protocol. The proposed study phases outlined in this amendment of the study protocol will include at least 200 qualifying subjects with intermittent suspension of the study to allow data analysis. The present study will continue until 200 CT positive test results (approximately 100 male and 100 female) are obtained. Of these 200 positive results, approximately 50% will be from symptomatic subjects and 50% from asymptomatic subjects. Since the positivity rate is presumably lower for asymptomatic subjects, the ration of symptomatic to asymptomatic subject enrollment for each study phase will be determined by the sponsor and will be made known in writing to each study site.

It is expected that approximately 3,000 subjects will be required to meet the overall study objectives. It is anticipated that the total number of subjects enrolled for testing throughout the study will yield approximately 30 positive NG samples (approximately 15 males and 15 females) with no requirement for a specific ratio of symptomatic to asymptomatic subjects. Subjects who are at high risk of exposure or suspect exposure to CT or NG, but are not currently being treated, will be recruited for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic females or males, age 14 or older, who present at a participating clinic with symptoms consistent with Chlamydia trachomatis or Neisseria gonorrhoeae infection, or
2. Asymptomatic females or males, age 14 or older, who present at a participating clinic and who suspect that they have CT and/or NG, or are considered at high risk of exposure (e.g., sexual partner that tests positive for CT, or NG, multiple sexual partners, ect.),
3. Individuals who are capable of understanding and agree to fulfill the requirements of the protocol.
4. Individuals who have signed the IRB approved informed consent form.

Exclusion Criteria:

1. Individuals with physical or mental inability that, in the opinion of the investigator can interfere with the subject's ability to follow the Identigene STD Test Collection Kit instructions,
2. Individuals who are currently being treated for CT or NG or who are currently receiving antibiotics or have received antibiotics within the last 28 days, and
3. Individuals who are suspected of being victims of sexual abuse or nonconsensual contact of a sexual nature within the previous 6 months or who are part of an ongoing sexual abuse legal case.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the Identigene STD Test Collection Kit in comparison to the Gen-Probe Aptima Combo 2 Assay | 1 day
  Demonstration of the effectiveness of the Identigene STD Test Collection Kit based on the percentage of concordant positive and negative results as compared to the Gen-Probe APTIMA Combo 2 assay conducted at an STD clinic.

SECONDARY OUTCOMES:
Evaluation of the Identigene STD Test Collection Kit instructions. | 1 day
  To determine if the instructions of the Identigene STD Test Collection Kit are adequate for proper specimen self-collection and specimen submission to the laboratory for processing.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Smith, Study Director — Lifetree Clinical Research; Lars Mouritsen, PhD, Study Chair — Identigene
Locations (1):
- John Hopkins University, Baltimore, Maryland, United States